CLINICAL TRIAL: NCT04380688
Title: A Phase 2, Open Label, Randomized Study of the Efficacy and Safety of Acalabrutinib With Best Supportive Care Versus Best Supportive Care in Subjects Hospitalized With COVID-19
Brief Title: Acalabrutinib Study With Best Supportive Care Versus Best Supportive Care in Subjects Hospitalized With COVID-19.
Acronym: CALAVI US
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Acerta Pharma BV (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D822FC00003
Record Dates: First submitted 2020-05-07; First posted 2020-05-08 (Actual); Results first posted 2021-09-13 (Actual); Last update posted 2021-09-13 (Actual); Status verified 2021-09

CONDITIONS: COVID-19
Keywords: 2019 novel coronavirus disease; Acalabrutinib; Btk inhibitor
MeSH Terms: conditions — COVID-19 | interventions — acalabrutinib

STUDY DESIGN:
Intervention Model Description: Study will consist of two arms Arm 1 is acalabrutinib + best supportive care or Arm 2 is best supportive care alone
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm 1 (Experimental): Acalabrutinib+ Best Supportive Care
  Interventions: Drug: Acalabrutinib
- Arm 2 (No Intervention): Best Supportive Care

INTERVENTIONS:
Drug: Acalabrutinib — Acalabrutinib administered orally
  Arms: Arm 1

SUMMARY:
CALAVI US will investigate the safety, efficacy and pharmacokinetics of acalabrutinib together with Best Supportive Care in the treatment of COVID-19.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to understand the purpose and risks of the study and provide signed and dated informed consent or have a legal representative provide consent and authorization to use protected health information (in accordance with national and local patient privacy regulations)
2. Men and women ≥18 years of age at the time of signing the informed consent form
3. Confirmed infection with SARS-CoV-2 confirmed per World Health Organization criteria (including positive RT-PCR nucleic acid test)
4. COVID-19 pneumonia (documented radiographically) requiring hospitalization and oxygen saturation <94% on room air or requires supplemental oxygen
5. Able to swallow pills
6. Willing to follow contraception guidelines

Exclusion Criteria:

1. Respiratory failure at the time of screening due to COVID-19 pneumonia that impedes the ability to swallow pills, or in the opinion of the treating physician, the subject is likely to require mechanical ventilation within the immediate 24 hours and therefore unable to swallow pills.
2. Known medical resuscitation within 14 days of randomization
3. Pregnant or breast feeding
4. Suspected uncontrolled active bacterial, fungal, viral, or other infection (besides infection with SARS-CoV-2)
5. Alanine aminotransferase (ALT), and/or aspartate aminotransferase (AST) and/or bilirubin ≥ 3x upper limit of normal (ULN) and/or severe hepatic impairment detected during the screening period (per local lab) Exception: AST and/or ALT ≤5 × ULN if considered due to underlying COVID-19 disease, but cannot be associated with concurrent elevated bilirubin (≤2 × ULN).
6. Uncontrolled or untreated symptomatic arrhythmias, myocardial infarction within the last 6 weeks, or congestive heart failure (NYHA Grade 3 or 4). Exception: Subjects with controlled, asymptomatic atrial fibrillation during screening are allowed to enroll
7. Treatment with a strong cytochrome P450 (CYP)3A inhibitor (within 7 days before first dose of study drug) or inducer (within 14 days before first dose of study drug).

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2020-06-13 (Actual); Primary Completion 2020-11-16 (Actual); Study Completion 2020-11-16 (Actual)

CONTACTS AND LOCATIONS:
Locations (28):
- United States (28):
  - Research Site, Anniston, Alabama
  - Research Site, Mobile, Alabama
  - Research Site, Escondido, California
  - Research Site, Fullerton, California
  - Research Site, Glendale, California
  - Research Site, Newport Beach, California
  - Research Site, New Haven, Connecticut
  - Research Site, Washington D.C., District of Columbia
  - Research Site, Fort Lauderdale, Florida
  - Research Site, Jacksonville, Florida
  - Research Site, Loxahatchee Groves, Florida
  - Research Site, Fort Wayne, Indiana
  - Research Site, Louisville, Kentucky
  - Research Site, Annapolis, Maryland
  - Research Site, Baltimore, Maryland
  - Research Site, Bethesda, Maryland
  - Research Site, Silver Spring, Maryland
  - Research Site, Hackensack, New Jersey
  - Research Site, Albany, New York
  - Research Site, Buffalo, New York
  - Research Site, New York, New York
  - Research Site, The Bronx, New York
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Nashville, Tennessee
  - Research Site, Houston, Texas
  - Research Site, Tyler, Texas
  - Research Site, Richmond, Virginia
  - Research Site, Renton, Washington

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal.
  All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the deidentified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- [Derived] Scheinberg P, Khoshnevis MR, Robinson PA, Guerreros A, Sato VAH, Fonseca BAL, Prozesky HW, Romero JOC, Fogliatto L, Meisenberg BR, Park DJ, Gupta A, Patel P, Townsley DM, Zheng L, Munugalavadla V. Efficacy and safety of acalabrutinib with best supportive care versus best supportive care in patients with COVID-19 requiring hospitalization. Immunohorizons. 2025 May 30;9(7):vlaf023. doi: 10.1093/immhor/vlaf023. PMID 40461100
- See also: Redacted CSP — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D822FC00003&attachmentIdentifier=2e2e7dff-ea3b-4994-b0b5-18b8ddb61ccb&fileName=D822FC00003_CSP_redacted.pdf&versionIdentifier=
- See also: Related Info — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D822FC00003&attachmentIdentifier=78253301-fe32-48e6-9d6a-56c0d83a543f&fileName=d822fc00003_SAP_redacted.pdf&versionIdentifier=
- See also: CSR Synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D822FC00003&attachmentIdentifier=fc178d1a-11fc-4fab-a215-d5459a97728f&fileName=D822FC00003_CSR_Synopsis_redacted.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All participants were recruited from the United States and had COVID-19 pneumonia (documented radiographically) requiring hospitalization. The first participant was randomized on 13 June 2020 and the last participant was randomized on 20 August 2020.
Pre-assignment Details: Screening assessments were performed within the 3 days prior to randomization. Of 70 screened participants, 62 were enrolled. Of the 8 participants that were not enrolled, 7 were screen failures (did not meet eligibility criteria) and 1 withdrew consent.
Groups:
- Acalabrutinib + BSC: Participants received acalabrutinib 100mg tablet orally twice daily for 10 days, plus best supportive care per the discretion of the Investigator and institutional guidelines.
- BSC Alone: Participants received best supportive care per the discretion of the Investigator and institutional guidelines.
Period: Overall Study
Arm/Group | Acalabrutinib + BSC | BSC Alone
Started | 31 | 31
Completed | 24 | 22
Not Completed | 7 | 9
Not completed — Death | 2 | 2
Not completed — Lost to Follow-up | 2 | 4
Not completed — Withdrawal by Subject | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Acalabrutinib + BSC | BSC Alone | Total
Number analyzed (Participants) | 31 | 31 | 62
Age, Continuous [Mean (Standard Deviation); unit: Years] | 52.5 (13.3) | 51.9 (14.3) | 52.2 (13.7)
Age, Customized [Number; unit: Participants]
  < 65 years | 26 | 25 | 51
  >= 65 years | 5 | 6 | 11
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 9 | 22
  Male | 18 | 22 | 40
Race/Ethnicity, Customized [Number; unit: Participants]
  HISPANIC OR LATINO | 15 | 13 | 28
  NOT HISPANIC OR LATINO | 16 | 17 | 33
  NOT REPORTED | 0 | 0 | 0
  MISSING | 0 | 1 | 1
Race/Ethnicity, Customized [Number; unit: Participants]
  WHITE | 18 | 20 | 38
  BLACK OR AFRICAN AMERICAN | 7 | 5 | 12
  AMERICAN INDIAN OR ALASKA NATIVE | 1 | 0 | 1
  ASIAN | 0 | 0 | 0
  NATIVE HAWAIIAN OR OTHER PACIFIC ISLANDER | 0 | 0 | 0
  OTHER | 3 | 2 | 5
  NOT REPORTED | 2 | 3 | 5
  MISSING | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events and Serious Adverse Events
Time Frame: Screening to 28 (+3) days after last dose of acalabrutinib (for acalabrutinib + BSC participants) or to 38 (+3) days after randomization (for BSC alone participants)
Population: Safety analysis set: If the participant receives at least 1 dose of acalabrutinib, they are summarized in the Acalabrutinib + BSC group. Otherwise, they are summarized in the BSC alone group.
  The number of participants in the BSC alone group (32) is greater than the number of participants randomized to this group (31) because one participant randomized to Acalabrutinib + BSC did not receive any acalabrutinib and therefore is included in the BSC alone group for the safety analysis set.
Measure: Count of Participants; unit: Participants
Arm/Group | Acalabrutinib + BSC | BSC Alone
Number analyzed (Participants) | 30 | 32
Participants
  Any Adverse Event | 17 | 15
  Any Serious Adverse Event | 4 | 6

2. Primary Outcome: Percentage of Participants Alive and Free of Respiratory Failure at Day 28
Description: Respiratory failure, is defined based on resource utilization of any of the following modalities: a) Endotracheal intubation and mechanical ventilation b) Oxygen delivered by highflow nasal cannula (heated, humidified, oxygen delivered via reinforced nasal cannula at flow rates >20 L/min with fraction of delivered oxygen ≥0.5) c) Noninvasive positive pressure ventilation or continuous positive airway pressure d) Extracorporeal membrane oxygenation
Time Frame: At Day 28
Population: Full analysis set (as randomized).
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | Acalabrutinib + BSC | BSC Alone
Number analyzed (Participants) | 31 | 31
Percentage of participants | 80.6 [67.4 to 93.9] | 83.9 [71.4 to 96.3]

3. Secondary Outcome: Percentage of Participants Alive and Free of Respiratory Failure at Day 14
Description: as for outcome 2
Time Frame: At Day 14
Population: Full analysis set (as randomized).
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | Acalabrutinib + BSC | BSC Alone
Number analyzed (Participants) | 31 | 31
Percentage of participants | 80.6 [67.4 to 93.9] | 87.1 [75.6 to 98.6]

4. Secondary Outcome: Percent Change From Baseline in C-reactive Protein.
Description: Baseline is defined as the result obtained on the date of randomization. If no result was obtained on the date of randomization, the last result prior to the date of randomization is used.
  Percent change from baseline at Day X is calculated by multiplying the following result by 100%: (Day X value - Baseline value)/Baseline value.
  The mean of this result for all analyzed patients is taken to get the mean percent change from baseline.
Time Frame: Days 3, 5, 7, 10, 14, 28
Population: Full analysis set (as randomized).
  Participants require a baseline and post-baseline result at the given timepoint to be included in the number analyzed for that timepoint.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Acalabrutinib + BSC | BSC Alone
Number analyzed (Participants) | 31 | 31
Percent change
  Day 3: number analyzed (Participants) | 27 | 24
  Day 3 | -41.08 (71.27) | -26.74 (69.02)
  Day 5: number analyzed (Participants) | 18 | 18
  Day 5 | -72.05 (26.29) | -49.55 (54.97)
  Day 7: number analyzed (Participants) | 11 | 12
  Day 7 | -75.72 (29.48) | -40.53 (75.99)
  Day 10/ Discharge (last post-baseline assessment if discharged from hospital prior to Day 10): number analyzed (Participants) | 30 | 29
  Day 10/ Discharge (last post-baseline assessment if discharged from hospital prior to Day 10) | -73.85 (27.92) | 9.23 (354.21)
  Day 10: number analyzed (Participants) | 5 | 7
  Day 10 | -73.23 (29.34) | 212.22 (710.39)
  Day 14: number analyzed (Participants) | 21 | 19
  Day 14 | -56.62 (97.54) | -56.61 (59.19)
  Day 28: number analyzed (Participants) | 19 | 14
  Day 28 | -66.89 (73.45) | -39.63 (161.97)

5. Secondary Outcome: Percent Change From Baseline in Ferritin
Description: as for outcome 4
Time Frame: Days 3, 5, 7, 10, 14, 28
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Acalabrutinib + BSC | BSC Alone
Number analyzed (Participants) | 31 | 31
Percent change
  Day 3: number analyzed (Participants) | 25 | 19
  Day 3 | -15.25 (21.87) | -7.38 (31.17)
  Day 5: number analyzed (Participants) | 14 | 12
  Day 5 | -29.67 (25.79) | -17.93 (36.74)
  Day 7: number analyzed (Participants) | 10 | 8
  Day 7 | -36.59 (22.78) | -9.67 (45.84)
  Day 10/ Discharge (last post-baseline assessment if discharged from hospital prior to Day 10): number analyzed (Participants) | 29 | 25
  Day 10/ Discharge (last post-baseline assessment if discharged from hospital prior to Day 10) | -24.48 (31.30) | -20.38 (28.00)
  Day 10: number analyzed (Participants) | 4 | 7
  Day 10 | -47.58 (31.60) | -1.24 (34.52)
  Day 14: number analyzed (Participants) | 19 | 18
  Day 14 | -45.25 (23.09) | -40.20 (26.81)
  Day 28: number analyzed (Participants) | 18 | 15
  Day 28 | -62.28 (37.27) | -63.69 (16.43)

6. Secondary Outcome: Percent Change From Baseline in Absolute Lymphocyte Count
Description: as for outcome 4
Time Frame: Days 3, 5, 7, 10, 14, 28
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Acalabrutinib + BSC | BSC Alone
Number analyzed (Participants) | 31 | 31
Percent change
  Day 3: number analyzed (Participants) | 17 | 17
  Day 3 | 54.75 (92.83) | 34.66 (61.47)
  Day 5: number analyzed (Participants) | 9 | 12
  Day 5 | 28.18 (64.35) | 76.86 (63.02)
  Day 7: number analyzed (Participants) | 6 | 9
  Day 7 | 46.22 (72.11) | 102.80 (107.71)
  Day 10/ Discharge (last post-baseline assessment if discharged from hospital prior to Day 10): number analyzed (Participants) | 19 | 20
  Day 10/ Discharge (last post-baseline assessment if discharged from hospital prior to Day 10) | 100.79 (142.10) | 97.45 (92.75)
  Day 10: number analyzed (Participants) | 3 | 6
  Day 10 | 67.41 (73.04) | 118.26 (66.81)
  Day 14: number analyzed (Participants) | 14 | 13
  Day 14 | 108.55 (110.73) | 106.85 (103.52)
  Day 28: number analyzed (Participants) | 11 | 11
  Day 28 | 135.30 (88.00) | 127.09 (136.57)

7. Secondary Outcome: Overall Survival
Description: Median overall survival, calculated using the Kaplan-Meier technique. Confidence interval for median overall survival (days) is derived based on Brookmeyer-Crowley method with log-log transformation.
Time Frame: From randomization until 90 days after randomization.
Population: Full analysis set (as randomized).
Measure: Median (90% Confidence Interval); unit: Days
Arm/Group | Acalabrutinib + BSC | BSC Alone
Number analyzed (Participants) | 31 | 31
Days | NA [NA to NA] — The median and lower and upper limit of the 95% confidence interval (CI) could not be calculated as there were an insufficient number of participants with events. | NA [NA to NA] — The median and lower and upper limit of the 95% confidence interval (CI) could not be calculated as there were an insufficient number of participants with events.

8. Secondary Outcome: Percentage of Participants Alive and Discharged From ICU
Time Frame: At Day 14 and at Day 28
Population: Full analysis set (as randomized).
Measure: Number; unit: Percentage of participants
Arm/Group | Acalabrutinib + BSC | BSC Alone
Number analyzed (Participants) | 31 | 31
Percentage of participants
  At Day 14 | 83.9 | 87.1
  At Day 28 | 83.9 | 87.1

9. Secondary Outcome: Time From Randomization to First Occurrence of Respiratory Failure or Death on Study Due to Any Cause
Description: Median time to first occurrence of respiratory failure or death, calculated using the Kaplan-Meier technique. Confidence interval for median overall survival (days) is derived based on Brookmeyer-Crowley method with log-log transformation.
Time Frame: From randomization to 28 days after randomization.
Population: Full analysis set (as randomized).
Measure: Median (90% Confidence Interval); unit: Days
Arm/Group | Acalabrutinib + BSC | BSC Alone
Number analyzed (Participants) | 31 | 31
Days | NA [NA to NA] — The median and lower and upper limit of the 95% confidence interval (CI) could not be calculated as there were an insufficient number of participants with events. | NA [NA to NA] — The median and lower and upper limit of the 95% confidence interval (CI) could not be calculated as there were an insufficient number of participants with events.
Statistical Analysis 1: Comparison: Acalabrutinib + BSC vs BSC Alone; Test type: Other — No formal hypothesis testing for this endpoint; Regression, Cox — P-value not generated; Adjusting for age (<65 vs >=65 years) and comorbidities (present vs absent). Ties handled by Efron approach. HR CI using profile likelihood approach; Hazard Ratio (HR) = 0.553, 90% CI 2-sided [0.145 to 1.952]

10. Secondary Outcome: Number of Days Alive and Free of Respiratory Failure
Description: as for outcome 2
Time Frame: From randomization to 28 days after randomization.
Population: Full analysis set (as randomized).
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Acalabrutinib + BSC | BSC Alone
Number analyzed (Participants) | 31 | 31
Days | 26.2 (6.7) | 24.6 (7.3)

11. Secondary Outcome: Number of Days With Respiratory Failure
Description: Respiratory failure, is defined based on resource utilization of any of the following modalities: a) Endotracheal intubation and mechanical ventilation b) Oxygen delivered by highflow nasal cannula (heated, humidified, oxygen delivered via reinforced nasal cannula at flow rates >20 L/min with fraction of delivered oxygen ≥0.5) c) Noninvasive positive pressure ventilation or continuous positive airway pressure d) Extracorporeal membrane oxygenation For participants who die (due to any cause) prior to Day 28, days from death to Day 28 are counted as days with respiratory failure. For participants in hospital and experiencing respiratory failure at the time they withdraw from the study, days from last known status to Day 28 are counted as days with respiratory failure.
Time Frame: From randomization to 28 days after randomization.
Population: Full analysis set (as randomized).
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Acalabrutinib + BSC | BSC Alone
Number analyzed (Participants) | 31 | 31
Days | 1.8 (6.7) | 3.4 (7.3)

12. Secondary Outcome: Number of Days Hospitalized
Description: For this summary, the hospitalization must be considered clinically indicated to count as a day hospitalized.
  For participants who die (due to any cause) prior to Day 28, days from death to Day 28 are counted as days hospitalized.
  For participants in hospital at the time they withdraw from the study, days from last known status to Day 28 are counted as days hospitalized.
Time Frame: From randomization to 28 days after randomization.
Population: Full analysis set (as randomized).
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Acalabrutinib + BSC | BSC Alone
Number analyzed (Participants) | 31 | 31
Days | 7.6 (7.3) | 9.0 (8.5)

13. Secondary Outcome: Number of Days in ICU
Description: For this summary, the ICU stay must be considered clinically indicated to count as a day in ICU.
  For participants who die (due to any cause) prior to Day 90, days from death to Day 90 are counted as days in ICU.
Time Frame: From randomization to 90 days after randomization.
Population: Full analysis set (as randomized).
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Acalabrutinib + BSC | BSC Alone
Number analyzed (Participants) | 31 | 31
Days | 4.4 (17.1) | 7.0 (20.8)

14. Secondary Outcome: Number of Days Alive Outside of Hospital
Time Frame: From randomization to 28 days after randomization.
Population: Full analysis set (as randomized).
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Acalabrutinib + BSC | BSC Alone
Number analyzed (Participants) | 31 | 31
Days | 20.2 (7.3) | 18.9 (8.6)

15. Secondary Outcome: Number of Days Alive Outside of Hospital
Time Frame: From randomization to 90 days after randomization.
Population: Full analysis set (as randomized).
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Acalabrutinib + BSC | BSC Alone
Number analyzed (Participants) | 31 | 31
Days | 75.3 (25.2) | 72.7 (25.0)

16. Secondary Outcome: Percent Change From Baseline in Oxygenation Index
Description: Baseline is defined as the result obtained on the date of randomization.
  Percent change from baseline at Day X is calculated by multiplying the following result by 100%: (Day X value - Baseline value)/Baseline value.
  The mean of this result for all analyzed patients is taken to get the mean percent change from baseline.
Time Frame: Days 3, 5, 7, 10, 14, 28
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Acalabrutinib + BSC | BSC Alone
Number analyzed (Participants) | 31 | 31
Percent change
  Day 3: number analyzed (Participants) | 28 | 26
  Day 3 | 14.24 (43.64) | 13.51 (30.67)
  Day 5: number analyzed (Participants) | 16 | 18
  Day 5 | 40.25 (74.37) | 18.71 (32.17)
  Day 7: number analyzed (Participants) | 12 | 12
  Day 7 | 18.41 (26.19) | 28.73 (31.15)
  Day 10/ Discharge (last post-baseline assessment if discharged from hospital prior to Day 10): number analyzed (Participants) | 30 | 30
  Day 10/ Discharge (last post-baseline assessment if discharged from hospital prior to Day 10) | 32.37 (66.33) | 36.67 (39.33)
  Day 10: number analyzed (Participants) | 4 | 9
  Day 10 | -23.81 (27.53) | 33.09 (50.42)
  Day 14: number analyzed (Participants) | 19 | 18
  Day 14 | 54.87 (84.54) | 59.22 (43.22)
  Day 28: number analyzed (Participants) | 18 | 18
  Day 28 | 48.87 (51.77) | 65.59 (50.76)

17. Secondary Outcome: Time From Randomization to Clinical Improvement of at Least 2 Points on a 9-point Category Ordinal Scale
Description: 9-point category ordinal scale: 0. * Uninfected, no clinical or virological evidence of infection
  1. Ambulatory, no limitation of activities
  2. Ambulatory, limitation of activities
  3. Hospitalized - mild disease, no oxygen therapy
  4. Hospitalized - mild disease, oxygen by mask or nasal prongs
  5. Hospitalized - severe disease, non-invasive ventilation or high flow oxygen
  6. Hospitalised - severe disease, intubation and mechanical ventilation
  7. Hospitalized - severe disease, ventilation and additional organ support, such as pressors, renal replacement therapy, extracorporeal membrane oxygenation
  8. Death
  Median time to first occurrence of respiratory failure or death, calculated using the Kaplan-Meier technique. Confidence interval for median overall survival (days) is derived based on Brookmeyer-Crowley method with log-log transformation.
Time Frame: From randomization to 28 days after randomization.
Population: Full analysis set (as randomized).
  Participants require a baseline and at least one post-baseline result to be included in the number analyzed.
Measure: Median (90% Confidence Interval); unit: Days
Arm/Group | Acalabrutinib + BSC | BSC Alone
Number analyzed (Participants) | 31 | 29
Days | 6.00 [5.00 to 7.00] | 7.00 [5.00 to 11.00]
Statistical Analysis 1: Comparison: Acalabrutinib + BSC vs BSC Alone; Test type: Other — No formal hypothesis testing for this endpoint; Regression, Cox — P-value not generated; [statistical method as in outcome 9, analysis 1]; Hazard Ratio (HR) = 1.314, 90% CI 2-sided [0.794 to 2.183]

18. Secondary Outcome: Pharmacokinetics of Acalabrutinib
Description: Summary of plasma concentrations (ng/mL) of acalabrutinib
Time Frame: Day 3 and Day 7
Population: PK analysis set: all participants who received at least 1 dose of acalabrutinib and had at least 1 post-dose evaluable pharmacokinetic (PK) data point for acalabrutinib or ACP-5862.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Acalabrutinib + BSC
Number analyzed (Participants) | 30
ng/mL
  Day 3, Pre-dose: number analyzed (Participants) | 8
  Day 3, Pre-dose | 6.258 (248)
  Day 3, 0.5 hours post-dose: number analyzed (Participants) | 14
  Day 3, 0.5 hours post-dose | 26.683 (173)
  Day 3, 1 hour post-dose: number analyzed (Participants) | 10
  Day 3, 1 hour post-dose | 210.858 (71.5)
  Day 3, 2 hours post-dose: number analyzed (Participants) | 18
  Day 3, 2 hours post-dose | 124.143 (89.2)
  Day 3, 4 hours post-dose: number analyzed (Participants) | 10
  Day 3, 4 hours post-dose | 33.714 (93.4)
  Day 7, 1 hour post-dose: number analyzed (Participants) | 1
  Day 7, 1 hour post-dose | 165.080 (NA) — Only 1 participant had a result for this timepoint.
  Day 7, 2 hours post-dose: number analyzed (Participants) | 0
  Day 7, 4 hours post-dose: number analyzed (Participants) | 1
  Day 7, 4 hours post-dose | 14.320 (NA) — Only 1 participant had a result for this timepoint.

19. Secondary Outcome: Pharmacokinetics of ACP-5862
Description: Summary of plasma concentrations (ng/mL) of ACP-5862
Time Frame: Day 3 and Day 7
Population: as for outcome 18
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Acalabrutinib + BSC
Number analyzed (Participants) | 30
ng/mL
  Day 3, Pre-dose: number analyzed (Participants) | 9
  Day 3, Pre-dose | 53.818 (140)
  Day 3, 0.5 hours post-dose: number analyzed (Participants) | 14
  Day 3, 0.5 hours post-dose | 58.959 (129)
  Day 3, 1 hour post-dose: number analyzed (Participants) | 10
  Day 3, 1 hour post-dose | 293.606 (68.1)
  Day 3, 2 hours post-dose: number analyzed (Participants) | 18
  Day 3, 2 hours post-dose | 273.528 (50.2)
  Day 3, 4 hours post-dose: number analyzed (Participants) | 10
  Day 3, 4 hours post-dose | 178.575 (44.2)
  Day 7, 1 hour post-dose: number analyzed (Participants) | 1
  Day 7, 1 hour post-dose | 582.180 (NA) — Only 1 participant had a result for this timepoint.
  Day 7, 2 hours post-dose: number analyzed (Participants) | 0
  Day 7, 4 hours post-dose: number analyzed (Participants) | 1
  Day 7, 4 hours post-dose | 139.560 (NA) — Only 1 participant had a result for this timepoint.

ADVERSE EVENTS:
Time Frame: Screening to 28 (+3) days after last dose of acalabrutinib (for acalabrutinib + BSC treated participants) or to 38 (+3) days after randomization (for BSC alone treated participants)
Description: Population summarized is the safety analysis set (treatment actually received): All participants who received at least 1 dose of acalabrutinib were included in Acalabrutinib + BSC arm, and patients who did not receive any acalabrutinib were included in BSC alone arm.
Arm/Group | Acalabrutinib + BSC | BSC Alone
All-Cause Mortality (participants affected / at risk) | 2/30 | 2/32
Serious Adverse Events (participants affected / at risk) | 4/30 | 6/32
Other Adverse Events (participants affected / at risk) | 5/30 | 3/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Acalabrutinib + BSC (N=30) | BSC Alone (N=32)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Retroperitoneal haematoma (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hepatotoxicity (Hepatobiliary disorders) | 1 (1) | 0 (0)
Portal vein thrombosis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Pneumonia cytomegaloviral (Infections and infestations) | 1 (1) | 0 (0)
Staphylococcal sepsis (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 2 (2)
Haemoglobin decreased (Investigations) | 0 (0) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 1 (1) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Acalabrutinib + BSC (N=30) | BSC Alone (N=32)
Headache (Nervous system disorders) | 4 (4) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 3 (3)

LIMITATIONS AND CAVEATS:
Improvements in BSC (use of corticosteroids and antivirals) have led to a substantial reduction in mortality and morbidity in patients hospitalized with COVID-19, which, in turn, minimizes the impact that additional treatment regimens can have on patient prognosis and recovery. In addition, variability in patient population and the performance of BSC across the globe poses challenges to demonstrate benefit.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI shall provide copies of any materials relating to the Study, or the Developed Technologies that either intends to publish or make any presentations relating to, at least 30 days in advance of publication, submission or presentation.

PI shall not include in or shall remove from any proposed publication of any Confidential Information, errors or inaccuracies; and shall withhold publication, submission for publication or presentation for 90 days from the date the Company receives the material.

DOCUMENTS (2):
  • Study Protocol (2020-07-24): https://cdn.clinicaltrials.gov/large-docs/88/NCT04380688/Prot_002.pdf
  • Statistical Analysis Plan (2020-10-01): https://cdn.clinicaltrials.gov/large-docs/88/NCT04380688/SAP_003.pdf